CLINICAL TRIAL: NCT07291583
Title: Clinical and Aesthetic Evaluation of Hyaluronic Acid in Addition to Connective Tissue Grafts in the Treatment of Gingival Recession Defects
Brief Title: Hyaluronic Acid With Connective Tissue Grafting for Gingival Recession
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Şeyma Çardakçı, asst. professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seyma9319
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - CTG + Hyaluronic Acid (Experimental): A 0.8% hyaluronic acid (HA) gel is applied to the connective tissue graft (CTG) before flap closure during the coronally advanced flap (CAF) procedure. The HA gel is used as an adjunctive biologic material to potentially enhance wound healing, soft tissue thickness, esthetic outcomes, and overall root coverage performance.
  Interventions: Biological: Hyaluronic Acid (0.8%) - Applied over CTG before flap closure (Test group only).; Procedure: Connective Tissue Graft + Coronally Advanced Flap (CTG + CAF)
- CTG only (Active Comparator): A standardized coronally advanced flap (CAF) procedure combined with a subepithelial connective tissue graft (CTG) is performed to treat gingival recession defects. The surgical protocol includes flap elevation, graft harvesting and placement, and flap advancement and suturing.
  Interventions: Procedure: Connective Tissue Graft + Coronally Advanced Flap (CTG + CAF)

INTERVENTIONS:
Biological: Hyaluronic Acid (0.8%) - Applied over CTG before flap closure (Test group only). — A 0.8% hyaluronic acid (HA) gel is applied to the connective tissue graft (CTG) before flap closure during the coronally advanced flap (CAF) procedure. The HA gel is used as an adjunctive biologic material to potentially enhance wound healing, soft tissue thickness, esthetic outcomes, and overall root coverage performance
  Arms: Experimental - CTG + Hyaluronic Acid
Procedure: Connective Tissue Graft + Coronally Advanced Flap (CTG + CAF) — A standardized coronally advanced flap (CAF) procedure combined with a subepithelial connective tissue graft (CTG) is performed to treat gingival recession defects. The surgical protocol includes flap elevation, graft harvesting and placement, and flap advancement and suturing.

SUMMARY:
This study evaluates whether adding 0.8% hyaluronic acid (HA) to connective tissue grafting and coronally advanced flap surgery improves clinical and esthetic outcomes in the treatment of gingival recession. Adult patients with Miller I-II or Cairo RT1 recession defects will be randomly assigned to receive CTG alone or CTG with adjunctive HA. Mean root coverage at 6 months is the primary outcome, while secondary measures include gingival thickness, clinical attachment level, esthetic scores, postoperative morbidity, and quality of life. The study aims to determine whether HA enhances soft tissue healing and root coverage predictability compared with conventional CTG.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least one gingival recession defect classified as Cairo RT1 or Miller Class I-II with a minimum depth of 1 mm.
* Full-mouth plaque score (FMPS) and full-mouth bleeding on probing (FMBOP) < 15%.
* Detectable cemento-enamel junction (CEJ).
* Age ≥ 18 years.
* No history of prior periodontal surgical treatment.
* Sufficient mental capacity to understand the study aims and procedures explained verbally and in writing.
* Determined to be cooperative and compliant with the clinician before, during, and after the surgical procedure.

Exclusion Criteria:

* Patients younger than 18 years.
* Periodontally healthy individuals.
* Current smokers.
* History of periodontal treatment within the past 1 year.
* Use of antibiotics within the past 3 months.
* Pregnancy or breastfeeding.
* Presence of systemic diseases such as diabetes, chronic kidney failure, cancer, bleeding disorders, connective tissue diseases, or other chronic conditions; and gingival recessions classified as Cairo RT3.
* Presence of cervical caries or restorations at the defect site.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Adjunctive Hyaluronic Acid on Mean Root Coverage After Recession Treatment | From enrollment to the end of treatment at 6 months"
  The primary objective of this study is to evaluate the effect of adjunctive hyaluronic acid (HA) on the mean root coverage (MRC) achieved after the treatment of gingival recession defects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gülhane Faculty of Dentistry, Ankara, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided